CLINICAL TRIAL: NCT01667107
Title: A Pharmacokinetic Analysis of Posaconazole in the Plasma and Alveolar Compartment of Lung Transplant Recipients
Brief Title: A Pharmacokinetic Analysis of Posaconazole in Lung Transplant Recipients (MK-5592-105)
Acronym: PAPAL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to an unfavorable risk-benefit analysis
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5592-105; 2012-003140-68 (EudraCT Number)
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posaconazole - CF Participants (Experimental): Posaconazole 400 mg oral solution twice daily administered with Calogen® to optimize absorption for a total of 6 weeks starting within 12 hours of leaving surgery, thereafter administered in the hospital or as an outpatient; the dose could be changed to posaconazole 200 mg 4 times per day if the participant is unable to meet the conditions for optimal absorption of posaconazole.
  Interventions: Drug: Posaconazole; Drug: Calogen®
- Posaconazole - Non-CF Participants (Experimental): Posaconazole 400 mg oral solution twice daily administered with Calogen® to optimize absorption for a total of 6 weeks starting within 12 hours of leaving surgery, thereafter administered in the hospital or as an outpatient; the dose could be changed to posaconazole 200 mg 4 times per day if the participant is unable to meet the conditions for optimal absorption of posaconazole.
  Interventions: Drug: Posaconazole; Drug: Calogen®

INTERVENTIONS:
Drug: Posaconazole
  Other Names: SCH056592; MK-5592; Noxafil®
Drug: Calogen®

SUMMARY:
This single site study will examine plasma and alveolar compartment (AC) levels of posaconazole in cystic fibrosis (CF) and non-cystic fibrosis (non-CF) lung transplant recipients receiving routine post-operative anti-fungal prophylaxis. Invasive fungal infection rates will be assessed following transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo lung transplantation
* Able to take oral/nasogastric medication
* Females of childbearing potential, males, and the sexual partners of males must use an effective method of birth control during this study and for 6 weeks after completing the study.

Exclusion Criteria:

* Severe liver disease
* Current use of cytochrome P-450 (CYP)-3A4 inhibitors including terfenadine, astemizole, cisapride, pimozide, halofantrine or quinidine within 7 days before transplant
* Treatment with posaconazole within 14 days before transplant
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01-23 (Actual); Primary Completion 2014-01-16 (Actual); Study Completion 2014-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=5592-105&kw=5592-105&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Cystic Fibrosis Participants: Cystic fibrosis participants received posaconazole 400 mg oral solution twice daily administered with Calogen® to optimize absorption for a total of 6 weeks starting within 12 hours of leaving surgery, thereafter administered in the hospital or as an outpatient; the dose could be changed to posaconazole 200 mg 4 times per day if the participant is unable to meet the conditions for optimal absorption of posaconazole.
- Non-Cystic Fibrosis Participants: Non-cystic fibrosis participants received posaconazole 400 mg oral solution twice daily administered with Calogen® to optimize absorption for a total of 6 weeks starting within 12 hours of leaving surgery, thereafter administered in the hospital or as an outpatient; the dose could be changed to posaconazole 200 mg 4 times per day if the participant is unable to meet the conditions for optimal absorption of posaconazole.
Period: Overall Study
Arm/Group | Cystic Fibrosis Participants | Non-Cystic Fibrosis Participants
Started | 8 | 18
Completed | 4 | 11
Not Completed | 4 | 7
Not completed — Adverse Event | 4 | 3
Not completed — Tolerability issues | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cystic Fibrosis Participants | Non-Cystic Fibrosis Participants | Total
Number analyzed (Participants) | 8 | 18 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.0 (7.82) | 52.4 (10.39) | 45.5 (14.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 3 | 11 | 14

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach 90% of the Steady State Serum Concentration of Posaconazole
Description: Blood samples for measurement of serum posaconazole were collected approximately 4 hours after the first daily dose on Days 1-12 and every Monday and Thursday on Days 13-43. The time to reach 90% of the steady state serum posaconazole concentration was to be estimated from fitting a linear model to the concentration data over time. The data did not permit estimation of the endpoint from the modeling proposed in the protocol.
Time Frame: Four hours after the first daily dose on Days 1-12 and every Monday and Thursday on Days 13-43
Population: The population to be analyzed included participants who complied with the protocol sufficiently to ensure that the results would exhibit the effects of treatment
Arm/Group | Cystic Fibrosis Participants | Non-Cystic Fibrosis Participants
Number analyzed (Participants) | 0 | 0

2. Post Hoc Outcome: Time to Reach a Serum Concentration of Posaconazole of >=0.5 mg/L
Description: Blood samples for measurement of serum posaconazole were collected approximately 4 hours after the first daily dose on Days 1-12 and every Monday and Thursday on Days 13-43. A posaconazole concentration >=0.5 mg/L is the therapeutic level, the concentration thought to lead to antifungal efficacy. The time at which the serum posaconazole concentration reached >=0.5 mg/mL and remained at that level for all subsequent assessments was recorded.
Time Frame: Four hours after the first daily dose on Days 1-12 and every Monday and Thursday on Days 13-43
Population: The population analyzed included all enrolled participants who reached and maintained posaconazole concentration of >=0.5 mg/L
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cystic Fibrosis Participants | Non-Cystic Fibrosis Participants
Number analyzed (Participants) | 6 | 14
Days | 12.2 (8.82) | 11.9 (9.86)

3. Post Hoc Outcome: Maximum Serum Concentration of Posaconazole (Cmax)
Description: Blood samples for measurement of serum posaconazole were collected approximately 4 hours after the first daily dose on Days 1-12 and every Monday and Thursday on Days 13-43. The maximum serum concentration of posaconazole was recorded.
Time Frame: Four hours after the first daily dose on Days 1-12 and every Monday and Thursday on Days 13-43
Population: The population analyzed included all enrolled participants
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cystic Fibrosis Participants | Non-Cystic Fibrosis Participants
Number analyzed (Participants) | 8 | 18
mg/L | 1.481 (0.6014) | 1.539 (0.8471)

4. Post Hoc Outcome: Time to Maximum Serum Concentration of Posaconazole (Tmax)
Description: Blood samples for measurement of serum posaconazole were collected approximately 4 hours after the first daily dose on Days 1-12 and every Monday and Thursday on Days 13-43. The time required to achieve the maximum serum concentration of posaconazole was recorded.
Time Frame: Four hours after the first daily dose on Days 1-12 and every Monday and Thursday on Days 13-43
Population: The population analyzed included all enrolled participants
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cystic Fibrosis Participants | Non-Cystic Fibrosis Participants
Number analyzed (Participants) | 8 | 18
Days | 19.5 (12.39) | 23.1 (13.73)

5. Primary Outcome: Concentration of Posaconazole in Bronchoalveolar Lavage (BAL) and Serum
Description: Concurrent BAL and serum samples for measurement of posaconazole concentration were to be collected during any clinically-indicated bronchoscopy. A participant could have more than 1 bronchoscopy.
Time Frame: Up to Day 42
Population: The population analyzed included all enrolled participants who had BAL and serum samples collected at the time of bronchoscopy and analyzed for posaconazole concentration. A participant could have more than 1 pair of samples (BAL and serum) included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/L
Units Other Than Participants: paired BAL and serum samples
Arm/Group | Cystic Fibrosis Participants | Non-Cystic Fibrosis Participants
Number analyzed (Participants) | 5 | 7
Number analyzed (paired BAL and serum samples) | 9 | 11
mg/L
  BAL | 1.116 (1.1699) | 0.764 (0.800)
  Serum | 0.829 (0.3742) | 0.7488 (0.3131)
Statistical Analysis 1: Comparison: Cystic Fibrosis Participants; Spearman rank correlation between concurrent BAL and serum posaconazole concentrations; Test type: Superiority or Other; p = 0.139, Spearman rank correlation; Spearman rank correlation coefficient = 0.53
Statistical Analysis 2: Comparison: Non-Cystic Fibrosis Participants; Spearman rank correlation between concurrent BAL and serum posaconazole concentrations; Test type: Superiority or Other; p = 0.057, Spearman rank correlation; Spearman rank correlation coefficient = 0.59

6. Secondary Outcome: Percentage of Participants Who Develop Invasive Fungal Infection
Description: Invasive fungal infection was assessed using the Mycoses Study Group/European Organisation for Research and Treatment of Cancer (MSG/EORTC) criteria. Infections counted in the analysis were those classified as 'proven', 'probable', or 'possible' according to the criteria.
Time Frame: Up to Day 84
Population: Participants were analyzed according to the group in which they were enrolled
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cystic Fibrosis Participants | Non-Cystic Fibrosis Participants
Number analyzed (Participants) | 8 | 18
Percentage of participants | 12.5 [2.2 to 47.1] | 16.7 [5.8 to 39.2]

ADVERSE EVENTS:
Time Frame: Up to Day 88
Description: All enrolled participants were assessed for adverse events. Adverse events that were serious and/or related to study drug were collected in the study. Related adverse events were those classified as possibly, probably, or certainly related to study drug.
Arm/Group | Cystic Fibrosis Participants | Non-Cystic Fibrosis Participants
Serious Adverse Events (participants affected / at risk) | 6/8 | 10/18
Other Adverse Events (participants affected / at risk) | 1/8 | 2/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cystic Fibrosis Participants (N=8) | Non-Cystic Fibrosis Participants (N=18)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Immunosuppressant drug level decreased (Investigations) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cystic Fibrosis Participants (N=8) | Non-Cystic Fibrosis Participants (N=18)
Nausea (Gastrointestinal disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Immunosuppressant drug level increased (Investigations) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation.